CLINICAL TRIAL: NCT01537822
Title: The Hysteroscopic Morcellator Versus the Bipolar Resectoscope for Removal of Lager Intrauterine Polyps, Removal of Submucous Myomas and Removal of Residual Placental Tissue: a Randomized Controlled Trial.
Brief Title: The Hysteroscopic Morcellator (HM).
Acronym: HM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/679
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2019-10

CONDITIONS: Large Intrauterine Polyps; Smaller Type 0 and 1 Myomas; Residual Placental Tissue
Keywords: intrauterine polyps; myomas; residual placental tissue
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- hysteroscopic morcellator (Experimental): Women, randomized into getting a treatment with the hysteroscopic morcellator.
  Interventions: Procedure: Hysteroscopic morcellator
- Resectoscope (Active Comparator): Women, randomized into getting a treatment with the resectoscope.
  Interventions: Procedure: Resectoscope

INTERVENTIONS:
Procedure: Hysteroscopic morcellator — Morcellation will be performed with the HM (TRUCLEAR, Smith & Nephew, Andover, USA). The rotary blade is used for polypectomy and removal of residual placental tissue; the reciprocating blade is used for myomectomy. The blade has a window-opening at the end with cutting edges through which tissue is aspirated by means of a vacuum source. The removed tissue is discharged through the device, collected in a pouch and made available for pathology analysis.
  Arms: hysteroscopic morcellator
Procedure: Resectoscope — Resectoscopy will be performed with a rigid 8.5 mm bipolar resectoscope (Karl Storz GmbH, Tuttlingen, Germany), equipped with a 0 or 30 degree optic. Normal saline is used for distension and irrigation of the uterine cavity. Fluid balance is closely monitored using a Hystero pump (Richard Wolf GmbH, Knittlingen, Germany) or Hysteromat pump (Karl Storz GmbH, Tuttlingen, Germany).
  Arms: Resectoscope

SUMMARY:
Rationale:

The hysteroscopic morcellator (HM) is a novel technique for removal of intrauterine polyps, myomas and placental tissue. It withholds some technical advantages over resectoscopy. Previous data suggest that it's a faster technique than the latter, and shows that it has a low complication rate.

Objective:

To compare the HM to bipolar resectoscopy for removal of:

1) large intrauterine polyps, 2) smaller type 0 and 1 myomas, 3) residual placental tissue, in terms of efficiency and complications.

Study design: Single blind, randomized controlled multicenter trial.

Study population: Women aged over 18 years old with:

1) large (≥ 1 cm) intrauterine polyps, 2) smaller (≤ 3 cm) type 0 or 1 myomas, 3) residual placental tissue, who are planned for hysteroscopic removal.

Intervention:

Patients are randomized between removal with the HM or the bipolar resectoscope.

Main study parameters/endpoints:

Installation and operating time.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Women who are referred to our polyclinic will be seen on a first visit, and, according to the standard work-up, an ultrasound will be performed when intrauterine pathology is suspected. To confirm the diagnosis a saline infusion sonography (SIS) and/or ambulant diagnostic hysteroscopy will be performed consequently. Once the diagnosis is confirmed and surgery is planned, women will be asked whether they want to take part in this study. At this moment, both techniques are used in our hospitals and the choice of treatment depends on the preference of the gynaecologist. All women will be treated with operative hysteroscopy in a daycare setting according to the standard of care, only now randomized between the two techniques. A standard postoperative visit with ultrasound examination and/or ambulant diagnostic hysteroscopy is scheduled 6 weeks later. Late postoperative complications and complaints are recorded.

It is expected that the HM beholds some advantages over the bipolar resectoscope such as shorter operating time and less complications (e.g. risk of perforation, current and fluid related complications). Previous data do not demonstrate any additional risks related to the use of the HM. Moreover we will check whether the HM has a lower risk of intrauterine adhesion formation, as this might influence patient's fertility.

After completion of the RCT, an observational study is planned considering pregnancies subsequent to the hysteroscopic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more intrauterine polyp(s) with a diameter ≥ 1 cm as seen on ultrasound, confirmed by saline infusion sonography and/or ambulant diagnostic hysteroscopy who are planned for hysteroscopic surgery.
* Patients with one or more intrauterine myoma(s) with a diameter ≤ 3 cm as seen on ultrasound, confirmed by saline infusion sonography and/or ambulant diagnostic hysteroscopy who are planned for hysteroscopic surgery.
* Patients with residual placental tissue as seen by ambulant diagnostic hysteroscopy who are planned for hysteroscopic surgery.

Exclusion Criteria:

* Only polyps < 1cm (Note: intrauterine polyps < 1 cm are treated in an ambulatory setting).
* Myomas with a diameter > 3 cm (Note: Myomas > 3 cm are treated with resectoscopy)
* Type 2 myomas
* Visual or pathological (e.g. on biopsy) evidence of malignancy preoperatively or at the time of operation.
* Untreated cervical stenosis making safe access for operative hysteroscopy impossible as diagnosed preoperatively or at the time of operation.
* With a contra-indication for operative hysteroscopy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-05; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Installation time and operating time. | the length of the operation
  Installation time is defined as the time to set up the hysteroscopic instrumentation ready for use (time from start of setting up the instrumentation to start resection / morcellation).
  Operating time is defined as the time starting visual introduction of the hysteroscope until the time at which the procedure is completed and the hysteroscope is removed definitely.
  Times will be measured with a stop watch by a trained nurse.
Check for adhesions during follow-up. | After 6 weeks, during follow-up visit
  Ambulant diagnostic hysteroscopy is performed at 6 weeks postoperative follow-up.

SECONDARY OUTCOMES:
Fluid deficit | during the length of the operation
  Fluid deficit in both procedures is the result of subtracting the outflow volumes from the inflow volumes as measured by the pump.
complications and complaints | between operation until 6 weeks follow-up
  During the postoperative hospital stay blood samples looking for electrolyte imbalances will only be taken when excessive fluid absorption is suspected based on fluid deficit (> 2500 mL for normal saline) and/or clinical symptoms.
  At 6 weeks postoperatively a standard visit is scheduled. Complications and complaints are recorded, and ultrasound is performed.

OTHER OUTCOMES:
Pregnancy rate | between the hysteroscopic removal of residual placental tissue and the first clinical pregnancy up to 7 years of follow-up
  number of pregnancies / number of women wishing to conceive
Pregnancy outcome | the first pregnancy subsequent to the hysteroscopic removal of residual placental tissue up to 7 years of follow-up
  Pregnancy outcome (biochemical / EUG / miscarriage / fetal demise / live birth)
Pregnancy complication | the first pregnancy subsequent to the hysteroscopic removal of residual placental tissue up to 7 years of follow-up
  Pregnancy complication (vaginal blood loss / preterm contractions / PPROM / pregnancy induced hypertension / preeclampsia / eclampsia / uterine rupture)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weyers, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Ghent University Hospital, Ghent, Belgium
- Catharina Hospital Eindhoven, Eindhoven, Netherlands

REFERENCES:
- [Derived] Hamerlynck TW, Schoot BC, van Vliet HA, Weyers S. Removal of Endometrial Polyps: Hysteroscopic Morcellation versus Bipolar Resectoscopy, A Randomized Trial. J Minim Invasive Gynecol. 2015 Nov-Dec;22(7):1237-43. doi: 10.1016/j.jmig.2015.07.006. Epub 2015 Jul 17. PMID 26192235
- See also: Related Info — http://www.uzgent.be